CLINICAL TRIAL: NCT04559334
Title: Compassionate-Use of 4% T-EDTA Lock Solution for Central Venous Lines of Pediatric PN Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: There is a new randomized controlled study being coordinated at Cincinatti Children's Hospital (Paul Wales MD, Principal Investigator). Only patients enrolled in this compassionate use study can continue to participate and is closed to new patients.
Sponsor: Boston Children's Hospital (Other)
Collaborators: SterileCare Inc. (Industry)
Responsible Party: Principal Investigator, Mark Puder, Senior Associate, Department of Surgery. Professor of Surgery, Harvard Medical School, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-P00035952
Record Dates: First submitted 2020-09-10; First posted 2020-09-22 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Central Line Complication; Central Line-associated Bloodstream Infection (CLABSI)
Keywords: central venous catheter; CLABSI; catheter occlusion; vascular access device; catheter patency; intestinal failure; parenteral nutrition
MeSH Terms: conditions — Intestinal Failure; Hyperphagia

STUDY DESIGN:
Intervention Model Description: Assessment of the effect of treatment will be based on a compassionate use study of parenterally administered 4% T-EDTA lock solution (KiteLock™ 4% Sterile Catheter Lock Solution) to determine safety and preliminary efficacy in the prevention of (1) thrombolytic occlusions, (2) catheter breakage and (3) CLABSI events. Each patient will serves as their own control with the catheter history 12 months' prior for each patient pre KiteLock ™ use (i.e., breakages, occlusions, CLABSIs) being compared with KiteLock ™ experience.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- open label (Other): All participants will receive Tetrasodium EDTA Catheter Lock Solution (KiteLock™ 4% Sterile Catheter Lock Solution)
  Interventions: Device: Tetrasodium EDTA Catheter Lock Solution

INTERVENTIONS:
Device: Tetrasodium EDTA Catheter Lock Solution — KiteLock™ 4% Sterile Catheter Lock Solution is a single use, clear, colorless and sterile solution. It is free of preservatives, alcohol and latex and is non-pyrogenic. KiteLock™ 4% is an aqueous solution containing a mixture of edetate tetrasodium and edetate trisodium. The solution composition is equivalent to 28 mg/mL edetate. EDTA is a known chelator. This means it has an affinity for metals and elements such as calcium. As a primary mechanism of action, it acts as a space occupying solution to prevent blood from entering the tip of the catheter when the catheter is not in use. As a secondary mechanism of action, it acts as an in vitro anticoagulant. This dual action decreases the risk of clot formation, consequently thrombolytic occlusions and by extension decreases the risk of CLABSI.
  Other Names: KiteLock™ 4% Sterile Catheter Lock Solution

SUMMARY:
In this research study we want to learn more about a study drug, tetrasodium sodium EDTA (Kitelock™) for maintaining the patency (blood flow) through a central venous catheter. Catheter occlusions such as blood clots have been shown to increase the risk of central line-associated bloodstream infection (CLABSI). This treatment consists of instilling a daily a dose of a solution , similar to heparin or saline lock flushes, into the catheter when it is not in use. The aim is to prevent CLABSI without increasing complications such as catheter breakage.

DETAILED DESCRIPTION:
Parenteral nutrition (PN) is a critical treatment for pediatric patients with intestinal failure (IF), defined as those unable to absorb nutrients enterally due to insufficient bowel length or function. Patients who require long term PN have an indwelling central venous line (CVL) for PN delivery. One risk of long-term PN use is the development of catheter occlusions and interruptions to device's patency. Such obstructions can lead to catheter breakage or embolization of the clot into the bloodstream, which can lead to stroke or death. Other complications related to long term use of indwelling CVLs are central line-associated bloodstream infection (CLABSI) and mechanical breakdown of the CVL. This is one of the most common complications of home PN. Among patients with a long-term CVL there are 250,000-500,000 episodes of CLABSI per year and among patients with CVLs for PN a range of 0.87-8.9 CLABSI episodes per 1000 catheter-days has been reported.

As stated, the development of CVL occlusions is a major risk associated with long term PN use. It occurs in as many as 25% of CVLs that are placed. Occlusion can be either partial or complete and has been defined as a decreased ability to infuse solutions into or withdraw solutions from a CVL. Occlusion can decrease flow rates, increase resistance and pressure, and potentially cause complete inability to withdraw and/or infuse fluid. Attempts at dissolving the occlusion may lead to catheter weakening or rupture due to the excessive pressure exerted on the device. Occlusions put a patient at further risk of morbidity and mortality due to delays in treatment and nutritional supplementation, or from fibrin deposition and resulting clot contributing to CLABSI. Additionally, the patient may have to undergo further invasive surgical interventions to replace the catheter.

Furthermore, the presence of occlusions within the CVL can predispose patients to CLABSIs as the clot can serve as reservoir for bacterial colonization. In some instances, the bacteria associated with the majority of CLABSIs are highly thrombogenic and create an environment suitable for the development additional thrombus. In patients with PN related cholestasis, sepsis is the biggest risk factor leading to the most common cause of death in these patients. Moreover, CLABSI is a major contributor to many other comorbidities (i.e., intestinal failure associated liver disease) and, when recurrent, has been recently shown to be a negative predictor in children who achieved enteral autonomy versus those who did not. CLABSI events are also a significant financial burden to both the patient and healthcare system and compromise to quality of life.

Locking solutions have been used in an effort to prevent CVL occlusions and CLABSIs with varying success. In the United States, saline and heparin have been used as the standard of care lock solution for decades. Both lock solutions however have fallen short of protecting patients against CVL complications and heparin has also caused serious systemic side effects as well as promoting biofilm formation within the lumen of CVLs. Compounded lock solutions such as taurolidine, citrate and ethanol and antibiotics have been used in the attempt to reduce CVL complications. Compounded 70% ethanol lock solutions have been used off label to eradicate organisms in biofilms present in CVLs and hence, treat or prevent CLABSIs. Ethanol also decreases the risk of antimicrobial resistance that may occur if concentrated antibiotic locks are used. Since the use of ethanol locks at Boston's Children Hospital (BCH) the CLABSI rate in IF patients dropped from 9.9 to 2.1 per 1000 catheter-days and reduced our morbidity and mortality. Unfortunately ethanol locks may alter the integrity of selected catheter materials, resulting in catheter breakage and leaching of the plasticizer into the bloodstream and frequent catheter occlusions. One meta analysis raised questions about the effect of the ethanol lock on catheter integrity based on the noted increase in catheter repair rates. Moreover, the currently available supply of sterile ethanol that is used to compound the locks has become prohibitively expensive. Homecare companies and retail pharmacies may no longer be able to provide them and it would be a significant out of pocket expense for patients and families if they had to pay for them. This lack of a reliable and affordable source of ethanol for CVL's places these vulnerable patients at a much higher risk of CLABSI and the associated morbidity and mortality.

Tetrasodium EDTA Catheter Lock Solution (KiteLock™ 4% Sterile Catheter Lock Solution) is produced by SterileCare Inc (Markham, Ontario, Canada) as a first generation product that focuses on reducing CVL complications. This 4% Tetrasodium EDTA (T-EDTA) solution is a dilution of EDTA in sterile water for injection. It was approved by Health Canada in 2016 as a Class II Medical Device, with Canada being the first market in the world to utilize it. It has subsequently received Canadian approval for use in children in July 2019. It is also currently approved for adult and pediatric use in Europe (CE mark) and Australia.

4% Tetrasodium-EDTA lock solution is known to improve catheter patency by working as an in vitro anticoagulant with in vitro antimicrobial activity against biofilm-forming Gram positive and negative bacteria, fungi and yeast. KiteLock™ 4% does not contribute to antibiotic resistance and does not contain any preservative, antibiotics, ethanol or latex. At the Toronto's Children Hospital in Canada, KiteLock™ 4% has been used since 2017 in their home PN population with previous history of line infections. Since its first approval in Canada, the use of 4% T-EDTA lock solution has been associated with a significant decrease in both catheter occlusions and CLABSI rates in CVLs of adult and pediatric PN patients.

Considering the growing concern with the lack of a reliable and affordable source of sterile ethanol injection, it is of the utmost importance to find a safe and effective replacement lock solution that will protect CVL lines against complications to avoid preventable emergency room visits at the hospital.

Therefore, based on a positive benefit-risk assessment taking into account its mechanisms of action and prior use children in Canada, KiteLock™ 4% is considered a potential lock replacement for the ethanol lock solution in pediatric PN patients followed by the Center for Advanced Intestinal Rehabilitation (CAIR) program at BCH. By following a Compassionate-Use Protocol, selected high-risk PN patients at BCH will be locking their CVLs daily with KiteLock™ 4%, and careful monitoring and follow-up for 12 months will determine the new lock's safety and efficacy in this patient population. These findings will be compared to each patient's previous catheter history 12 months' prior while receiving ethanol lock; in other words, each subject will serve as their own control.

1. Specific Aims /Objectives

1.1 To determine the safety and efficacy profile of 4% T-EDTA lock solution (KiteLock™ 4% Sterile Catheter Lock Solution) acting to maintain catheter patency and thus prevent thrombotic occlusions and related complications.

1.2 To determine whether the pattern of catheter occlusions and catheter breakage in patients receiving 4% T-EDTA lock solution is different than what was experienced when they were previously receiving the compounded 70% ethanol lock solution.

Secondary Aims To determine whether the pattern of CLABSIs in patients receiving 4% T-EDTA lock solution is different than what was experienced when they were previously receiving the compounded 70% ethanol lock solution.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a tunneled central venous catheter or peripherally inserted central catheter (PICC) for administration of PN or intravenous hydration fluids to treat intestinal failure
2. Patients aged 3 months to 18 years old inclusive
3. Minimum patient weight of at least 5 kilograms
4. History of at least one thrombolytic occlusion and/or CLABSI event
5. Signed patient informed consent
6. Clinically stable for at least 4 weeks with no acute medical co-morbidities

Exclusion Criteria:

1. Pregnancy or nursing mother
2. Enrollment in any other clinical trial involving an investigational agent (unless approved by the principal investigators of the other trial)
3. The parent or guardian or child unwilling to provide consent or assent
4. Clinical instability such as the following:

   * Acute pulmonary edema
   * Acute myocardial infarction
   * Acute stroke
   * Acute thromboembolism
   * Metabolic acidosis
   * Sepsis
   * Coagulopathy with prolonged activated partial thromboplastin time (aPTT) or international normalized ratio (INR)
   * Severe hypoglycemia
5. Subjects who are hypersensitive or allergic to EDTA
6. Active therapy with long-term anti-microbial agents, such as taurolidine (not including patients receiving intermittent antimicrobial treatment for small intestinal bacterial overgrowth)
7. A compromised catheter defined as one which has been repaired several times.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Number of participants with Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | through study completion, an average of 1 year
  The number of treatment-related events as assessed by CTCAE v4.0 will be tracked for all study participants receiving 4% T-EDTA lock solution
The Number of Participants with Catheter Occlusions | through study completion, an average of 1 year
  The number of participants with catheter occlusions based on thrombolytic usage or need for catheter removal as assessed during clinical visits and admissions to the hospital or emergency room.
The Number of Participants with Catheter Breaks | through study completion, an average of 1 year
  The number of catheter breaks requiring catheters to be repaired or replaced will be collected based on emergency room and hospital records.

SECONDARY OUTCOMES:
The Number of Central Line Associated Bloodstream Infections (CLABSIs) | through study completion, an average of 1 year
  The number and pattern CLABSIs in participants will be assessed based on emergency room and hospital records.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Puder, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Childrens's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the the study, the results will be published in a peer reviewed journal - including incidence of catheter occlusions, catheter breaks, and CLABSI events.
  Upon request we will share study protocol and supporting materials (consent, how to obtain device)
Supporting Information: Study Protocol, ICF
Time Frame: To be determined.
Access Criteria: To be determined.

REFERENCES:
- [Background] Hirsch TI, Fligor SC, Tsikis ST, Mitchell PD, DeVietro A, Carbeau S, Wang SZ, McClelland J, Carey AN, Gura KM, Puder M. Administration of 4% tetrasodium EDTA lock solution and central venous catheter complications in high-risk pediatric patients with intestinal failure: A retrospective cohort study. JPEN J Parenter Enteral Nutr. 2024 Jul;48(5):624-632. doi: 10.1002/jpen.2644. Epub 2024 Jun 5. PMID 38837803
- [Background] Safdar N, Kluger DM, Maki DG. A review of risk factors for catheter-related bloodstream infection caused by percutaneously inserted, noncuffed central venous catheters: implications for preventive strategies. Medicine (Baltimore). 2002 Nov;81(6):466-79. doi: 10.1097/00005792-200211000-00007. PMID 12441903
- [Background] Clare A, Teubner A, Shaffer JL. What information should lead to a suspicion of catheter sepsis in HPN? Clin Nutr. 2008 Aug;27(4):552-6. doi: 10.1016/j.clnu.2008.04.013. Epub 2008 Jul 26. PMID 18662842
- [Background] Reimund JM, Arondel Y, Finck G, Zimmermann F, Duclos B, Baumann R. Catheter-related infection in patients on home parenteral nutrition: results of a prospective survey. Clin Nutr. 2002 Feb;21(1):33-8. doi: 10.1054/clnu.2001.0500. PMID 11884010
- [Background] Squires RH, Duggan C, Teitelbaum DH, Wales PW, Balint J, Venick R, Rhee S, Sudan D, Mercer D, Martinez JA, Carter BA, Soden J, Horslen S, Rudolph JA, Kocoshis S, Superina R, Lawlor S, Haller T, Kurs-Lasky M, Belle SH; Pediatric Intestinal Failure Consortium. Natural history of pediatric intestinal failure: initial report from the Pediatric Intestinal Failure Consortium. J Pediatr. 2012 Oct;161(4):723-8.e2. doi: 10.1016/j.jpeds.2012.03.062. Epub 2012 May 11. PMID 22578586
- [Background] Toure A, Duchamp A, Peraldi C, Barnoud D, Lauverjat M, Gelas P, Chambrier C. A comparative study of peripherally-inserted and Broviac catheter complications in home parenteral nutrition patients. Clin Nutr. 2015 Feb;34(1):49-52. doi: 10.1016/j.clnu.2013.12.017. Epub 2014 Jan 3. PMID 24439240
- [Background] Ross VM, Guenter P, Corrigan ML, Kovacevich D, Winkler MF, Resnick HE, Norris TL, Robinson L, Steiger E. Central venous catheter infections in home parenteral nutrition patients: Outcomes from Sustain: American Society for Parenteral and Enteral Nutrition's National Patient Registry for Nutrition Care. Am J Infect Control. 2016 Dec 1;44(12):1462-1468. doi: 10.1016/j.ajic.2016.06.028. PMID 27908433
- [Background] Chang MI, Carlson SJ, Nandivada P, O'Loughlin AA, Potemkin AK, Cowan E, Mitchell PD, Gura KM, Puder M. Challenging the 48-Hour Rule-Out for Central Line-Associated Bloodstream Infections in the Pediatric Intestinal Failure Population: A Retrospective Pilot Study. JPEN J Parenter Enteral Nutr. 2016 May;40(4):567-73. doi: 10.1177/0148607114567897. Epub 2015 Jan 7. PMID 25567785
- [Background] Stephens LC, Haire WD, Kotulak GD. Are clinical signs accurate indicators of the cause of central venous catheter occlusion? JPEN J Parenter Enteral Nutr. 1995 Jan-Feb;19(1):75-9. doi: 10.1177/014860719501900175. PMID 7658605
- [Background] Mehall JR, Saltzman DA, Jackson RJ, Smith SD. Fibrin sheath enhances central venous catheter infection. Crit Care Med. 2002 Apr;30(4):908-12. doi: 10.1097/00003246-200204000-00033. PMID 11940768
- [Background] Crowley AL, Peterson GE, Benjamin DK Jr, Rimmer SH, Todd C, Cabell CH, Reller LB, Ryan T, Corey GR, Fowler VG Jr. Venous thrombosis in patients with short- and long-term central venous catheter-associated Staphylococcus aureus bacteremia. Crit Care Med. 2008 Feb;36(2):385-90. doi: 10.1097/01.CCM.0B013E3181611F914. PMID 18091541
- [Background] Raad II, Luna M, Khalil SA, Costerton JW, Lam C, Bodey GP. The relationship between the thrombotic and infectious complications of central venous catheters. JAMA. 1994 Apr 6;271(13):1014-6. PMID 8139059
- [Background] Thornburg CD, Smith PB, Smithwick ML, Cotten CM, Benjamin DK Jr. Association between thrombosis and bloodstream infection in neonates with peripherally inserted catheters. Thromb Res. 2008;122(6):782-5. doi: 10.1016/j.thromres.2007.10.001. Epub 2007 Nov 13. PMID 17997477
- [Background] Timsit JF, Farkas JC, Boyer JM, Martin JB, Misset B, Renaud B, Carlet J. Central vein catheter-related thrombosis in intensive care patients: incidence, risks factors, and relationship with catheter-related sepsis. Chest. 1998 Jul;114(1):207-13. doi: 10.1378/chest.114.1.207. PMID 9674471
- [Background] Shanks RM, Donegan NP, Graber ML, Buckingham SE, Zegans ME, Cheung AL, O'Toole GA. Heparin stimulates Staphylococcus aureus biofilm formation. Infect Immun. 2005 Aug;73(8):4596-606. doi: 10.1128/IAI.73.8.4596-4606.2005. PMID 16040971
- [Background] Modi BP, Jaksic T. Pediatric intestinal failure and vascular access. Surg Clin North Am. 2012 Jun;92(3):729-43, x. doi: 10.1016/j.suc.2012.03.012. PMID 22595718
- [Background] Liu F, Hansra S, Crockford G, Koster W, Allan BJ, Blondeau JM, Lainesse C, White AP. Tetrasodium EDTA Is Effective at Eradicating Biofilms Formed by Clinically Relevant Microorganisms from Patients' Central Venous Catheters. mSphere. 2018 Nov 28;3(6):e00525-18. doi: 10.1128/mSphere.00525-18. PMID 30487154